CLINICAL TRIAL: NCT01638169
Title: The Contribution of Heels for Walking Quality Among Children With Muscular Dystrophy
Status: Completed | Type: Observational
Sponsor: Alyn Pediatric & Adolescent Rehabilitation Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 920100239
Record Dates: First submitted 2012-07-09; First posted 2012-07-11 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2015-06

CONDITIONS: Step Time and Length; Symmetry; Step Time and Length Variability; Heart Rate; Gait Velocity

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 20 children with DMD
  Interventions: Device: adding a heel

INTERVENTIONS:
Device: adding a heel — walking with and without heels on the gaitrite system

SUMMARY:
During the stand phase the DMD foot is too plantarflexed in addition patients adopt a higher flexion and abduction of the hip in order to advance the swinging limb. The aim of this work is to assess the immediate contribution of heels for these walking disturbance in children with muscular dystrophy disease.

ELIGIBILITY:
Inclusion Criteria:

* age >6 yrs
* walk without heel strike

Exclusion Criteria:

* cannot understand simple instructions

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children with DMD age >6 yrs walk without heel strike
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2013-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
gait parameters | pre and post heels adj.

CONTACTS AND LOCATIONS:
Locations (1):
- Alyn, Jerusalem, Israel